CLINICAL TRIAL: NCT03560661
Title: Identification of Acoustic and Perceptual Markers of Lower and Upper Motor Neuron Signs in Dysarthria of Patients With Amyotrophic Lateral Sclerosis : a Comparison With Primitive Lateral Sclerosis, Kennedy's Disease and Controls
Brief Title: Acoustic and Perceptual Markers of Dysarthria in Amyotrophic Lateral Sclerosis (ALS)
Acronym: SPEECH-ALS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: NI17040J; 2017-A03151-52 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-01-02; First posted 2018-06-18 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Kennedy's Disease
Keywords: Acoustic and perceptual markers; Dysarthria; Amyotrophic lateral sclerosis; Primitive lateral sclerosis; Kennedy's disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Bulbo-Spinal Atrophy, X-Linked; Dysarthria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amyotrophic lateral sclerosis (ALS) patients
- Primitive Lateral Sclerosis (PLS) patients
- Kennedy's disease (KD) patients

SUMMARY:
This study proposes to identify acoustic and perceptual markers related to upper motor neuron (UMN) degeneration and lower motor neuron (LMN) degeneration in the dysarthria of patients with amyotrophic lateral sclerosis (ALS) which involves the degeneration of both systems. ALS patients will be gathered in clinical groups according to electromyogram (EMG) and clinical signs observed in the bulbar site. UMN signs are defined as jaw clonus, gag reflex and pseudobulbar features (lability). LMN signs are defined as lingual atrophy and fasciculations. The dysarthria will be compared to dysarthria of patients involving an exclusive UMN system degeneration (in primitive lateral sclerosis) and an exclusive LMN system degeneration (Kennedy's disease). Patients will be compared to the controls who permitted to establish the standards of the "MonPaGe" tool. MonPaGe is a computerized tool based on a multidimensional and quantified assessment of voice and speech, by a set of targeted acoustic and perceptual criteria.

DETAILED DESCRIPTION:
ALS is a motor neuron disease characterized by a progressive degeneration of motor neurons in the brain, brainstem, and spinal cord. Degeneration of the upper and lower motor neurons (UMN and LMN) leads to spasticity, impaired reflexes, muscle fatigue, muscle weakness and atrophy. PLS is a motor neuron disease involving exclusively the UMN system and Kennedy's disease is a genetic condition involving the LMN system. Those three different motor neuron diseases can lead to a dysarthria. Affected individuals with ALS vary significantly in the locus of disease onset, presentation at diagnosis and rate of progression. Regardless of the site of onset, most patients with ALS will experience bulbar motor deterioration that will lead to a dysarthria. According to Darley's classification of dysarthrias, dysarthria in ALS is grossly described as "mixed" (both spastic, due the UMN deterioration, and flaccid, due to the LMN deterioration). However, at the onset of bulbar signs, when the dysarthria is still mild, dysarthric profiles and bulbar clinical signs can vary within individuals. Perceptual and acoustic features of dysarthria in ALS have been studied but they have not been studied in dysarthric patients with PLS and KD. This study was motivated by the need to better understand the dysarthria in ALS and it's management in speech therapy. The goals of this study is to question the impact of the degeneration of the UMN system versus the LMN system on the speech motor system and see if the investigators can identify acoustic and perceptual markers related to UMN degeneration on one side and LMN degeneration on the other side. The investigators will compare acoustic and perceptual features between the recorded speech of different clinical groups. Clinical groups will be made according to clinical signs and EMG. The clinical signs for UMN involvement in the bulbar region are: gag reflex, jaw clonus, pseudobulbar features (lability). The clinical signs for LMN involvement are: lingual atrophy and fasciculation. The population will be composed by groups of ALS-LMN patients, ALS-UMN patients , PLS patients and KD patients and a control group already recruited by the LPP (Laboratoire de Phonétique et de Phonologie) team (CNRS...) which permitted to establish the standards of the "MonPaGe" tool that the investigators will use to analyse patients recorded speech. This tool is based on a multidimensional and quantified assessment of voice and speech, by a set of targeted acoustic and perceptual criteria.

ELIGIBILITY:
Inclusion Criteria:

* Major patients diagnosed at the "centre référent des maladies du motoneurone" with ALS, PLS or KD,
* French motherhood language
* Mild to moderate severity of dysarthria according to the Perceptual Score of the BECD
* Without respiratory troubles according to the neurologist
* Without dementia.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 80 patients (40 ALS patients, 20 PLS patients and 20 KD patients). They will be recruited at the "centre de référence pour les maladies du motoneurone (Pitié-Salpêtrière). An initial EMG will be achieved during the usual diagnostic management
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Number of patients in each patterns of dysarthria | 1 day
  Patterns of dysarthria will be determined with post hoc unsupervised machine learning method (cluster analysis) from following measurements:
  * Intelligibility: number of words recognized (score 0 to 15)
  * Maximum phonation time (TMP), (milliseconds),
  * Phonation: mean and standard deviation of fundamental frequency (Hz); jitter (%), shimmer (%);Signal to Noise Ratio (dB)
  * Intensity modulation capacities (score 0 to 4),
  * Articulation of consonants and vowels : global error score (score 0 to 53); qualitative profile of error; acoustic range variation (Hz),
  * Coarticulation (Hz),
  * Score of prosody,
  * Verbal Diadococinesis : accuracy (score 0 to 4) ; control (score 0 to 4) and flow rate (syllables/sec),
  * Speech flow rate (syllables/sec).

SECONDARY OUTCOMES:
Functional scale with the Norris score | 1 day
  The functional capacities of the bulbar site will be evaluated by the speech therapist with the Norris score.This examination will permit to identify UMN and LMN signs
Functional scale with the ALS functional rating scale-R (ALS FRS-R) | 1 day
  The functional capacities of the bulbar site will be evaluated by the speech therapist with the ALS functional rating scale-R (ALS FRS-R). This examination will permit to identify UMN and LMN signs
Severity of the dysarthria | 1 day
  A severity score of the dysarthria will be calculated with the Perceptual Score of the Batterie d'Evaluation Clinique de la Dysarthrie (BECD)
Clinical examination | 1 day
  Classical speech therapy clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LEVEQUE, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- APHP - Hôpital Pitié-Salpêtriere, Paris, France

REFERENCES:
- [Derived] Slis A, Leveque N, Fougeron C, Pernon M, Assal F, Lancia L. Analysing spectral changes over time to identify articulatory impairments in dysarthria. J Acoust Soc Am. 2021 Feb;149(2):758. doi: 10.1121/10.0003332. PMID 33639779